CLINICAL TRIAL: NCT04813900
Title: Correlation Between Lung UltraSound Score and Hypoxemia for Interstitial Syndrome in Emergency Department
Acronym: O2LUSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Dupriez Florence, Principal investigator, MD Consultant in Emergency Medicine, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/10FEV/062
Record Dates: First submitted 2021-03-19; First posted 2021-03-24 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient suspected to suffer from interstitial syndrome needing an arterial blood gas analysis (Experimental)
  Interventions: Other: Lung ultrasound

INTERVENTIONS:
Other: Lung ultrasound — Lung ultrasound in order to calculate lung ultrasound score

SUMMARY:
The primary objective of this study is to assess the presence of a correlation between the Lung ultrasound score (LUSS) and PaO2/FiO2 in patient presenting with interstitial syndrome (IS) in the ED. The primary end point considers the null hypothesis to be a negative linear distribution for LUSS and PaO2/FiO2 values.

Secondary objectives and secondary end points One of the secondary objectives is to assess the correlation between the LUSS and PaCO2 in patient presenting with IS in the ED. The end point of this secondary outcome considers the null hypothesis to be a positive linear distribution for the LUSS and PaCO2 values.

Another secondary objective is to determine the influence of the presence of unilateral or bilateral pleural effusion on the correlation between LUSS and PaO2/FiO2. The end point of this secondary outcome considers the null hypothesis to be a negative linear distribution for LUSS and PaO2/FiO in those three sub-groups: absence of pleural effusion group, unilateral pleural effusion group and bilateral pleural effusion group.

DETAILED DESCRIPTION:
Justification for the research

Interstial lung disease (ILD) is characterized by a diffuse affection of the lung interstitial tissue. It can be secondary to acute conditions such as pneumonia or pulmonary oedema either of haemodynamic aetiology either permeability induced. ILD can also result from chronic diffuse parenchymal lung disease (DPLD). It is admitted that acute ILD leads to decreased pulmonary aeration and therefore to hypoxemia.

In front of a patient presenting in Emergency Department (ED) with altered oxygen saturation, arterial blood is classically sampled. Arterial Blood Gases (ABG) procedure, in addition to be painful for the patient, is invasive. ABG however gives access, among other results, to the Arterial Pressure in Oxygen (PaO2), which evaluates the level of hypoxemia. Although the correlation between ABG results and prognosis hasn't been widely evaluated, a rather recent study supported the absence of correlation between those for Acute Heart Failure (AHF). Authors however did not report the correlation between severity of symptoms at patient's hospital admission and hypoxemia. Yet, according to the Berlin definition, hypoxemia represented by the ratio PaO2/FiO2 is a severity indicator in Acute Respiratory Distress Syndrome (ARDS).

Lung ultrasound is a simple tool, non-invasive, non-irradiating, low cost and easily available at the patient's bedside. In addition, ultrasound equipment has become wildly available in the ED and more and more portable. Simultaneously, the interest of lung ultrasound for critically ill patient has been demonstrated. The ILD ultrasonographic diagnosis is based on the presence of multiple ultrasound artefacts called B-lines. B-lines appear when the ratio between air and water is abnormal. Different anatomic substrates have been recognized as being at the origin of this ultrasound pattern. In acute pulmonary oedema the presence of B-lines is related to the presence of extra-vascular water. B-lines presence is also attributed to the thickening of sub-pleural interlobular septa. B-lines are therefore a representation of ILD and accessible using ultrasound. Additionally, more and more ultrasound machines are provided with options to quantify the number of B-lines.

Regarding the importance of B-lines and their interconnection to ILD, a score has been created to evaluate ILD. The Lung Ultrasound Score (LUSS) is based on B-lines quantitative assessment. The B-lines detection is performed in six thoracic zones bilaterally. In each zone, ultrasound lung aeration status is determined scoring from zero to four. A normal aeration of the lung with presence of A lines, persistent pleural sliding and less than three B-lines scores zero point. An ILD, resulting in moderate loss of aeration with more than three spaced B-lines, 7mm apart, scores one point. An alveolar-interstitial syndrome meaning a severe loss of aeration with coalescent B-lines, less then 3mm apart, scores two. An alveolar consolidation leading to a complete loss of aeration with an ultrasonographic tissue like pattern, scores three. A total score over thirty-six can be calculated using this method. Initially developed on an experimental model resembling various pathological conditions encountered in the critically ill, LLUS proved to be correlated to the different states of aeration of the lung. Literature findings are consistent with LUSS being an efficient tool to measure lung aeration in different intensive care situations: re-aeration antibiotics-induced in Ventilator Associated Pneumonia, assessment of PEEP-induced lung recruitment. LUSS realized during weaning trial has been showed to be able to predict of post-extubation distress. In the Intensive Care Unit (ICU), LUSS is efficient to quantify lesions and predict mortality associated with ARDS.

Knowing LUSS has a good correlation to the lung aeration, the present physiological study is meant to highlight a potential negative linear correlation between PaO2/FiO2 values and LUSS. If this hypothesis is confirmed, the LUSS could eventually be a tooltool indirectly assessing the impact of an ILD on haematosis and correlating the potential degree of hypoxemia in the emergency room for patients with this acute pathology. This could secondary increase patient's comfort by reducing ABG realization for follow up.

Study procedure:

Intervention description

A LUSS will be realized by an investigator trained for lung ultrasound (LUS) and considering him/herself confident for its use. A five-point Likert scale will be filled. To the statement "I am qualified to realize a LUSS", only emergency doctors answering "I strongly agree" or "I agree" will be eligible for inclusion and added to investigators list using an amendment to this protocol. The ultrasound machines operated for LUS belong to each ED meaning the investigators are familiar to its use. To standardize the results, settings of the ultrasound machines will be standardized. To allow the exploration of the pulmonary parenchyma a low frequency curvilinear transducer will be used and evaluation of B-lines will be performed using a depth of at least 12cm as commonly recommended1. In this SARS-COV-2 pandemic context, patients affected with this condition having a pulmonary involvement could reach our eligibility criteria. Therefore, special precautions, such as a single protection cover of the ultrasound machine and proper use of disinfectant for probes will be recommended between patients. Those measures will follow institutional procedures of ultrasound use during COVID19 pandemic. LUS will take place within 10 minutes of ABG analysis. LUS will be performed at the patient's bedside. The investigator will be blinded to any other procedure made by treating physician for diagnostic purpose. The LUSS procedure will be used as validated for ARDS15. For that matter, the thorax is virtually divided in six thoracic zones bilaterally, comporting two anterior zones, two lateral zones and two posterior zones. The anterior and lateral zones will be evaluated in strict dorsal decubitus and the posterior zones will be evaluated with a light contro-lateral decubitus allowed, if necessary because of patient morphotype. For each zone a score from zero to three will be determined:

* 0: A normal aeration of the lung with presence of A lines, persistent pleural sliding and less than three B-lines.
* 1: Interstitial syndrome, resulting in moderate loss of aeration with more than three spaced B-lines, 7mm apart, scores one point.
* 2: Alveolar-interstitial syndrome meaning a severe loss of aeration with coalescent B-lines, less then 3mm apart, scores two.
* 3: An alveolar consolidation leading to a complete loss of aeration with an ultrasonographic tissue like pattern.

LUSS will be calculated by adding the score given to each 12 zones, with a maximum of thirty-six. Patients scoring less than two, will be considered empirically with no interstitial syndrome and will be secondary excluded of the study. Investigators will also report the presence of pleural effusion allowing to classify the patient in one of these three subgroups:

* Absence of pleural effusion
* Unilateral pleural effusion
* Bilateral pleural effusion In order to collect those results, a template with a reminder about how to calculate the LUSS will be joined to the Case Report Form (CRF). The result of LUSS won't be communicated to the treating physician.

Study conduction

The study flow chart is displayed in Figure 3.

Study Setting

Before the study launching, the investigator will be recruited using a five-point Likert scale as previously described. A presentation of the study and the procedure will be organized by the coordinating investigators in each including ED.

Patients' recruitment

The eligible patients will be identified by the treating ED physician. Patients admitted to ED with dyspnea, without taking account of any dyspnea classification, and for which the ED physician decide on the basis of his clinical judgment the realization of an ABG, will be considered for inclusion. The decision of the realization of an ABG being left to the ED physician, ABG is not considered as an intervention. Patients less than eighteen years old, patients presenting with a known chronic IS, COPD or patients for which LUS is not feasible will be discarded.

Inclusion

All eligible patients will undergo a LUSS after having given an informed consent to the investigator. The target population will include patients temporary not able to give a written and informed consent due to their acute condition. Therefore, the consent will either be written or verbal with secondary signature as soon as possible. Any legal representative will also be given the possibility to sign consent. Only patients with written consent will be included for data analysis. In Belgium, LUS isn't recognized as standard of care giving to this study an interventional character. The result of the LUSS will not be communicated to the treating physician.

Secondary exclusion Patients with a LUSS of less than 2 will not be considered as affected with IS and be secondary excluded.

Data collection and Data treatment

The LUSS will be reported on a template included in the CFR. It will be filled out by the investigator and joined to the signed consent. Name, first name, date of birth and hospital administrative number of the included patients will be recorded on the CFR. Investigators will only access personal data of the patient they have personally included; principal investigators will have access to all personal data in order to be able to collect missing data. Data will secondary be replaced by neutral identifier for analysis.

Follow up

There will be no follow up.

Statistics

The software IBM SPSS statistics 23.0 (SPSS Inc., Chicago, IL, USA) will be used to analyse our data. Since LUSS will be considered as a continuous value for all of our analysis, Pearson formula was used to calculate the patient sample. For the description of our population, the continuous values will be expressed in mean with a minimal and maximal values and standard deviations while discrete values will be reported by categories and expressed in numbers and percentage. Comparison between quantitative data will be realized with a Chi2-test and comparison between continuous data with a Wilcoxon-Mann-Whitney test. Significance threshold will be set with a p-value at <0.05. Confidence intervals will be 95% and calculate using " Mid-P exact value ".

Data Management

Data circuit and confidentiality

The paper CRFs will be collected in each centre by the principal investigators and hand-delivered to the study promoter. Patients will initially be identified on the CRF by their last name, first name, date of birth, file's number from the institution where they have been included and an identification's number from the study. This identification's number will include a reference for the inclusion centre, a number of inclusions, the first letter of the patient name and month and year of birth. After completion of the collection of missing data by principal investigators, patients will only be identified by their study identification number in order to be anonymised. A list of correspondence between study identification number and the other identifying data initially collected will be kept under the responsibility of the promoter. This list is kept for the statutory period of time provided for this type of research. The protection of the patient's personal data will be guaranteed according to the European General Data Protection Regulation of 27 April 2016 (in application since 25 May 2018), to the Belgian Law of 30 July 2018 on the protection of privacy with regard to the processing of personal data and to the Belgian Law of 22 August 2002 on the rights of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent
* >17 years old
* Arterial Blood Gas analysis at admission
* Lung ultrasound within 10 minutes of ABG sample

Exclusion Criteria:

* Patient with pathologies leading to chronic interstitial syndrome
* Chronic Obstructive Pulmonary Disease (COPD)
* Lung ultrasound not feasible: pneumonectomy history, severe obesity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the presence of a correlation between the LUSS and PaO2/FiO2 in patient presenting with IS in the ED | 6 months
  The primary end point considers the null hypothesis to be a negative linear distribution for LUSS and PaO2/FiO2 values.

SECONDARY OUTCOMES:
correlation between the LUSS and PaCO2 in patient presenting with IS in the ED | 6 months
  The end point of this secondary outcome considers the null hypothesis to be a positive linear distribution for the LUSS and PaCO2 values.
influence of the presence of unilateral or bilateral pleural effusion on the correlation between LUSS and PaO2/FiO2 | 6 months
  The end point of this secondary outcome considers the null hypothesis to be a negative linear distribution for LUSS and PaO2/FiO in those three sub-groups: absence of pleural effusion group, unilateral pleural effusion group and bilateral pleural effusion group

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires saint luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837
- [Result] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Result] Fan E, Brodie D, Slutsky AS. Acute Respiratory Distress Syndrome: Advances in Diagnosis and Treatment. JAMA. 2018 Feb 20;319(7):698-710. doi: 10.1001/jama.2017.21907. PMID 29466596
- [Result] Minana G, Nunez J, Banuls P, Sanchis J, Nunez E, Robles R, Mascarell B, Palau P, Chorro FJ, Llacer A. Prognostic implications of arterial blood gases in acute decompensated heart failure. Eur J Intern Med. 2011 Oct;22(5):489-94. doi: 10.1016/j.ejim.2011.01.014. Epub 2011 Feb 25. PMID 21925058
- [Result] Mojoli F, Bouhemad B, Mongodi S, Lichtenstein D. Lung Ultrasound for Critically Ill Patients. Am J Respir Crit Care Med. 2019 Mar 15;199(6):701-714. doi: 10.1164/rccm.201802-0236CI. PMID 30372119
- [Result] Lichtenstein D, Meziere G, Biderman P, Gepner A, Barre O. The comet-tail artifact. An ultrasound sign of alveolar-interstitial syndrome. Am J Respir Crit Care Med. 1997 Nov;156(5):1640-6. doi: 10.1164/ajrccm.156.5.96-07096. PMID 9372688
- [Result] Lichtenstein DA, Meziere GA, Lagoueyte JF, Biderman P, Goldstein I, Gepner A. A-lines and B-lines: lung ultrasound as a bedside tool for predicting pulmonary artery occlusion pressure in the critically ill. Chest. 2009 Oct;136(4):1014-1020. doi: 10.1378/chest.09-0001. PMID 19809049
- [Result] Soldati G, Copetti R, Sher S. Sonographic interstitial syndrome: the sound of lung water. J Ultrasound Med. 2009 Feb;28(2):163-74. doi: 10.7863/jum.2009.28.2.163. PMID 19168766
- [Result] Agricola E, Bove T, Oppizzi M, Marino G, Zangrillo A, Margonato A, Picano E. "Ultrasound comet-tail images": a marker of pulmonary edema: a comparative study with wedge pressure and extravascular lung water. Chest. 2005 May;127(5):1690-5. doi: 10.1378/chest.127.5.1690. PMID 15888847
- [Result] Jambrik Z, Monti S, Coppola V, Agricola E, Mottola G, Miniati M, Picano E. Usefulness of ultrasound lung comets as a nonradiologic sign of extravascular lung water. Am J Cardiol. 2004 May 15;93(10):1265-70. doi: 10.1016/j.amjcard.2004.02.012. PMID 15135701
- [Result] Bellani G, Rouby JJ, Constantin JM, Pesenti A. Looking closer at acute respiratory distress syndrome: the role of advanced imaging techniques. Curr Opin Crit Care. 2017 Feb;23(1):30-37. doi: 10.1097/MCC.0000000000000380. PMID 27906709
- [Result] Via G, Lichtenstein D, Mojoli F, Rodi G, Neri L, Storti E, Klersy C, Iotti G, Braschi A. Whole lung lavage: a unique model for ultrasound assessment of lung aeration changes. Intensive Care Med. 2010 Jun;36(6):999-1007. doi: 10.1007/s00134-010-1834-4. Epub 2010 Mar 11. PMID 20221746
- [Result] Bouhemad B, Liu ZH, Arbelot C, Zhang M, Ferarri F, Le-Guen M, Girard M, Lu Q, Rouby JJ. Ultrasound assessment of antibiotic-induced pulmonary reaeration in ventilator-associated pneumonia. Crit Care Med. 2010 Jan;38(1):84-92. doi: 10.1097/CCM.0b013e3181b08cdb. PMID 19633538
- [Result] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923
- [Result] Soummer A, Perbet S, Brisson H, Arbelot C, Constantin JM, Lu Q, Rouby JJ; Lung Ultrasound Study Group. Ultrasound assessment of lung aeration loss during a successful weaning trial predicts postextubation distress*. Crit Care Med. 2012 Jul;40(7):2064-72. doi: 10.1097/CCM.0b013e31824e68ae. PMID 22584759
- [Result] Zhao Z, Jiang L, Xi X, Jiang Q, Zhu B, Wang M, Xing J, Zhang D. Prognostic value of extravascular lung water assessed with lung ultrasound score by chest sonography in patients with acute respiratory distress syndrome. BMC Pulm Med. 2015 Aug 23;15:98. doi: 10.1186/s12890-015-0091-2. PMID 26298866